CLINICAL TRIAL: NCT03544112
Title: NIDA CTN-0079: Emergency Department Connection to Care With Buprenorphine for Opioid Use Disorder
Brief Title: Emergency Department Connection to Care With Buprenorphine for Opioid Use Disorder
Acronym: ED-CONNECT
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 17-01513
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ED and OUD treatment providers and staff: * ED patients will be recruited to participate in interviews or focus groups.
  * ED patients who are eligible for and willing to receive ED-initiated BUP will be recruited to participate in two research visits.
  * Administrative and health record data will be examined to assess rates of screening, assessment, eligibility determination, etc.
  Interventions: Behavioral: Employ a multifaceted approach to facilitate clinical protocol implementation
- Community Stakeholders: * Community treatment providers/OTP leadership and program staff: Providers, leadership and staff involved in the provision of office-based BUP, community treatment, and/or at opioid treatment programs (OTPs) will be recruited to participate in the formative evaluation and the Implementation Facilitation.
  * Other Stakeholders: Other community leaders and members (e.g., EMS, fire department, police, local government leadership, community advocacy groups, etc.) may be recruited to participate in qualitative interviews or focus groups.
  Interventions: Behavioral: Employ a multifaceted approach to facilitate clinical protocol implementation
- Patients: ED patients will be recruited to participate in interviews or focus groups.
  Interventions: Behavioral: Employ a multifaceted approach to facilitate clinical protocol implementation; Drug: Initiate BUP (SL-BUP or XR-BUP) in the ED

INTERVENTIONS:
Behavioral: Employ a multifaceted approach to facilitate clinical protocol implementation — Implementation will include developing clinical protocols containing core components of the intervention to which fidelity is expected, along with aspects that may be adapted by local sites to aid implementation. In partnership with multidisciplinary teams at each site, we will adapt clinical practices from other contexts and available information about SL-BUP and XR-BUP to site-specific clinical protocols and implementation strategies. The study implementation facilitators will assist local champions to identify potential treatment providers and draw on existing resources for training and ongoing support.
Drug: Initiate BUP (SL-BUP or XR-BUP) in the ED — The study implementation facilitators will assist local champions to identify potential treatment providers and draw on existing resources for training and ongoing support.
  Groups: Patients

SUMMARY:
The purpose of this study is to learn what resources are needed to improve outcomes for patients with opioid use disorder. The study will look at how patients engage in treatment and the decisions that patients and providers make regarding treatment, specifically buprenorphine treatment, for opioid use disorder.

The aims of this study are:

1. To evaluate using mixed methods the feasibility and acceptability of OUD screening, ED-initiated BUP, and referral.
2. Over the course of the study and as XR-BUP is added to hospital formularies, to estimate the percentage and confidence intervals of patients assessed, treated, and engaged in treatment at Day 30. This will be a three-site study employing a multi-faceted approach to facilitate clinical protocol implementation and to assess feasibility, acceptability, and impact. Investigators will develop, introduce and update site-specific ED clinical protocols and implementation plans for OUD screening, ED-initiated BUP, and referral for treatment. A participatory action research approach will be utilized along with mixed methods incorporating data derived from:

   * Medical record and administrative data abstraction,
   * Research assessments involving patients who are eligible for and willing to receive ED-initiated BUP (including both those who do, and do not, receive BUP); these assessments will document the index ED visit and the 30th day after the index ED visit,
   * Qualitative interviews, focus groups, and quantitative assessments involving providers and staff, patients, and other stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* ED STAFF: ED/Hospital leadership and staff: Leadership and staff across multiple disciplines (e.g., nurses, social workers, physicians, NPs, PAs, pharmacist, physician and nursing directors) at each ED site will be recruited to participate in the formative evaluation and the IF.
* PROVIDERS: Community treatment providers/OTP leadership and program staff: Providers, leadership and staff involved in the provision of office-based BUP, community treatment, and/or at opioid treatment programs (OTPs) will be recruited to participate in the formative evaluation and the Implementation Facilitation.
* COMMUNITY: Other Stakeholders: Other community leaders and members (e.g., EMS, fire department, police, local government leadership, community advocacy groups, etc.) may be recruited to participate in qualitative interviews or focus groups.
* PATIENTS: ED patients will be recruited to participate in interviews or focus groups.
* PATIENT-PARTICIPANTS: ED patients who are eligible for and willing to receive ED-initiated BUP will be recruited to participate in two research visits.
* ALL ED PATIENTS: Administrative and health record data will be examined to assess rates of screening, assessment, eligibility determination, etc.

Stakeholder-Participant Inclusion Criteria

* A member of one of the stakeholder groups (1-4 above)

Patient-Participant Inclusion Criteria

* Eligible for and willing to receive ED-initiated BUP

  1. Eligibility for ED-initiated BUP is operationally defined as meeting site clinical protocol criteria determined and documented by site clinical staff. See Section 9.2 Clinical Protocol.
  2. Willing to receive ED-initiated BUP is operationally defined as providing an affirmative answer to the following question, which will be embedded in each site's clinical protocol: Would you like to receive buprenorphine today?
  3. NOTE: Patients meeting these criteria, and not meeting exclusion criteria below, may be included as study participants regardless of whether they receive or do not receive ED-initiated BUP

Exclusion Criteria:

Stakeholder-Participant Exclusion Criteria

* Unwilling or unable to provide consent
* Currently in jail, prison or any inpatient overnight facility as required by court of law or have pending legal action or that could prevent participation in the study

Patient-Participant Exclusion Criteria

* Not able to speak English sufficiently to understand study procedures and provide written informed consent
* Unable or unwilling to provide written informed consent or to participate in study procedures
* Currently receiving any medication treatment for OUD at the time of index ED visit
* Current research participant in a substance use intervention study or previous participation in the current study
* Are currently in jail, prison or any inpatient overnight facility as required by court of law or have pending legal action or that could prevent participation in the study
* Inadequate locator information (unable to provide 2 unique means of contact)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a three-site study employing a multi-faceted approach to facilitate clinical protocol implementation and to assess feasibility, acceptability, and impact
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
Receipt of ED-initiated BUP (binary) and will be abstracted from the health record. | 12 Months
  Proportion receiving emergency department BUP amongst patients who have been determined to be eligible for and willing to receive ED-initiated BUP

SECONDARY OUTCOMES:
Proportion of patients who received ED-initiated BUP who are engaged in formal addiction treatment 30 days after the index ED visit. | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Ryan McCormack, MD, Principal Investigator — NYU Langone Health
Locations (4):
- United States (4):
  - Valley Regional Healthcare, Claremont, New Hampshire
  - Catholic Medical Center, Manchester, New Hampshire
  - Bellevue Hospital Center, New York, New York
  - New York University School of Medicine, New York, New York

REFERENCES:
- [Derived] McCormack RP, Rotrosen J, Gauthier P, D'Onofrio G, Fiellin DA, Marsch LA, Novo P, Liu D, Edelman EJ, Farkas S, Matthews AG, Mulatya C, Salazar D, Wolff J, Knight R, Goodman W, Williams J, Hawk K. Implementing Programs to Initiate Buprenorphine for Opioid Use Disorder Treatment in High-Need, Low-Resource Emergency Departments: A Nonrandomized Controlled Trial. Ann Emerg Med. 2023 Sep;82(3):272-287. doi: 10.1016/j.annemergmed.2023.02.013. Epub 2023 May 2. PMID 37140493
- [Derived] McCormack RP, Rotrosen J, Gauthier P, D'Onofrio G, Fiellin DA, Marsch LA, Novo P, Liu D, Edelman EJ, Farkas S, Matthews AG, Mulatya C, Salazar D, Wolff J, Knight R, Goodman W, Hawk K. Implementation facilitation to introduce and support emergency department-initiated buprenorphine for opioid use disorder in high need, low resource settings: protocol for multi-site implementation-feasibility study. Addict Sci Clin Pract. 2021 Mar 9;16(1):16. doi: 10.1186/s13722-021-00224-y. PMID 33750454